CLINICAL TRIAL: NCT07382206
Title: Effect of Acute Exercise on Sleep Patterns in Patients With PLMS Using a Wearable Device Compared With a Control Group
Brief Title: Effect of Acute Exercise on Sleep Patterns in Patients With PLMS, Using a Wearable Device, Compared With a Control Group ( SONEX )
Acronym: SONEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Samsung Eletrônica da Amazônia Ltda (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 84402424.5.0000.5599
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Periodic Leg Movements, Excessive, Sleep-Related
Keywords: Polysomnography; sleep; Device; Periodic Limb Movements of Sleep; Cardiopulmonary Exercise Test
MeSH Terms: conditions — Nocturnal Myoclonus Syndrome | interventions — Exercise Test; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Intervention Model Description: Effect of a single session of acute exercise on objective sleep patterns in adults with and without PLMS, as assessed by polysomnography. For this analysis, mobile and wearable devices will be employed to monitor physiological parameters that will serve as biomarkers of both exercise and sleep. In addition, study questionnaires will be administered, advanced glycation end-products (AGEs) will be evaluated, and participants will use the study devices (smartwatch and smart ring) at home for seven consecutive days.
Masking Description: Participants will be assigned to the PLM or control groups based on polysomnography results indicating the presence or absence of PLM events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLM Group (Experimental): A single session of acute intense exercise will influence sleep-related biological parameters assessed by polysomnography, including the number of PLMS events.
  Interventions: Procedure: Cardiopulmonary Exercise Test (CPET) - Twice
- Control Group (Experimental): A single acute session of intense exercise will be reflected in sleep biological parameters measured by polysomnography, including the number of PLMS events.
  Interventions: Procedure: cardiopulmonary exercise test (CPET)

INTERVENTIONS:
Procedure: cardiopulmonary exercise test (CPET) — The participant will perform a single session of acute exercise 4 hours prior to polysomnography. On the same day, shortly before the polysomnography, study questionnaires will be administered, and the study devices (watch and ring) will be placed on the participant to record electrophysiological sleep parameters in conjunction with the polysomnography. The following morning, participants will be discharged and will continue to use the devices and complete study questionnaires at home for seven consecutive days. After the seven-day period, participants will return to undergo the second and final polysomnography. On this day, prior to the polysomnography, participants will complete study questionnaires, and advanced glycation end-products (AGEs) will be measured using the AGEs device and the smartwatch.
  Arms: Control Group
Procedure: Cardiopulmonary Exercise Test (CPET) - Twice — The participant will undergo a single session of acute exercise (CPET) 4 hours prior to polysomnography (PSG). Before the PSG, study questionnaires will be administered, and the participant will wear study devices (smartwatch and smart ring) to collect sleep and physiological data during the night, in conjunction with the (PSG).
  The next day, participants will be discharged and begin a seven-day free-living period, during which they will continue using the devices at night. After this seven-day period, participants will return for a second PSG. On this day, prior to the PSG, participants will complete study questionnaires, and advanced glycation end-products (AGEs) will be measured using the AGE scanner device and the smartwatch. This description outlines the first block of the protocol.
  Following an interval of up to seven days to 3 weeks, the protocol will be repeated as described above, excluding the final PSG. This repetition constitutes the 2º block of the protocol.
  Arms: PLM Group

SUMMARY:
The effects of chronic exercise on health promotion, improvement of quality of life, and reduction of the risk of developing chronic diseases such as obesity, diabetes mellitus, cardiovascular diseases, depression, and cancer are well established. In addition, the positive influence of exercise on sleep patterns and sleep quality is widely recognized. However, few studies have addressed the effects of a single session of physical exercise on the circadian cycle and sleep disorders.

Regarding Periodic Limb Movement Disorder (PLMD), which is characterized by periodic episodes of repetitive and highly stereotyped limb movements, the scientific literature indicates that the effects of a single session of intense exercise remain insufficiently explored. Therefore, the present study aims to investigate, through a controlled interventional study, the effects of acute exercise on the Periodic Limb Movements of Sleep (PLMS) index.

To this end, the study will recruit healthy participants as well as individuals with PLMS to perform acute exercise sessions, followed by a polysomnographic examination and a longitudinal observation period. Throughout the study, participants will use wearable and mobile devices to monitor their physiological patterns. In addition, questionnaires related to sleep, physical exercise, cognitive decline, and depression will be administered to better characterize the study population.

Thus, this study aims to generate evidence regarding the influence of acute exercise on sleep patterns in participants with PLMS, as well as to obtain data to support the development of algorithms related to sleep quality, including PLMS detection, which may be embedded in wearable or mobile devices in the future.

ELIGIBILITY:
General Inclusion Criteria:

* Aged 22 years or older;
* Self-reported habitual sleep of at least 5 consecutive hours per night. Specific Inclusion Criteria for the PLMS Group
* Having a prior polysomnography (PSG) showing a PLMS index ≥ 15/h;
* Screening PSG for participants without a PSG in the last 6 months showing a PLMS index ≥ 15/h.

Note: Efforts will be made to ensure that approximately 50% of the sample consists of participants with a PLMS index > 50/h. -

General Exclusion Criteria:

* Pregnant or lactating individuals;
* Presence of dermatological conditions or skin diseases such as vitiligo, lupus, atopic dermatitis, or tattoos on the wrist or fingers that could interfere with optical sensor readings from the smartwatch or smart ring;
* Inability to attend the study PSG sessions;
* Use of medications indicated for the treatment of sleep disorders;
* Current or prior treatment for PLMS management;
* Presence of implanted cardiac devices, such as pacemakers, cardioverter defibrillators, or cardiac resynchronization devices;
* Prior diagnosis of chronic neurological, orthopedic, cardiac, pulmonary, or other clinical conditions that limit the ability to perform physical activity.

Specific Exclusion Criteria for the Control Group:

-Presence of sleep disorders identified on the screening PSG, such as: moderate to severe sleep apnea (apnea-hypopnea index [AHI] ≥ 15), insomnia with an Insomnia Severity Index (ISI) score above 14, or PLMS index > 15.-

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sleep parameters measured by polysomnography | 7 days
  A single acute session of intense exercise will be reflected in sleep-related biological parameters measured by polysomnography, including the number of PLMS events. Furthermore, the exercise effect will also be compared between two different groups: individuals with PLMS and those without PLMS.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Cristine Treptow, PhD, Principal Investigator — Instituto do Sono
Locations (1):
- CDEC Brasil, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The parties have agreed that the data will be shared with the study collaborator exclusively in anonymized form.